CLINICAL TRIAL: NCT00383604
Title: Breast Cancer Lymphedema: Role of Insulin Resistance/FOXC2
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: California Breast Cancer Research Program (Other)
Responsible Party: Sponsor
Other Study IDs: BRSNSTU0009; 96204 (Other: Stanford University Alternate IRB Approval Number); BRSNSTU0009 (Other: Stanford University); 2580 (Other: Stanford IRB)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Lymphedema; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To better understand the mechanisms leading to lymphedema development in breast cancer survivors, and the implications for potential innovative approaches to the screening, prevention and treatment of this condition.

DETAILED DESCRIPTION:
Lymphedema of the arm is an important, under-recognized, and under-treated complication of successful surgical and radiotherapeutic treatment of breast cancer. As a result of advances in early detection and effective adjuvant therapies, many women diagnosed with breast cancer today can expect survival that is similar to age-matched women without breast cancer. Nevertheless, this source of substantial physical and psychological morbidity has not attracted sufficient attention from industry or the scientific research community to result in either effective risk stratification or the availability highly effective therapeutic interventions.

While the presence and degree of arm edema can, in part, correlated with the extent of axillary surgery, we still comprehend only poorly the factors that predispose to overt lymphatic insufficiency in the patients at risk for lymphedema by virtue of prior breast cancer treatment. It is likely that this anatomic and regenerative variability relies, at least in part, upon an as yet undefined genetic substrate. A growing body of evidence suggests that mutations in the nuclear transcription gene FOXC2 are responsible for a broad clinical array of primary lymphedema syndromes. The biology of breast cancer-associated lymphedema, including its characteristic latency phase, suggests that similar mechanisms may operate in the predisposition to this and other forms of secondary lymphedema.

In parallel, breast cancer-associated lymphedema has several clinical attributes that suggest a relationship to, and a role for, insulin resistance. In this regard, it is interesting to contemplate the recent, multiple lines of evidence that suggest that the gene FOXC2 regulates, directly or indirectly, several aspects of adipocyte metabolism and that genetic variability in the gene may influence features associated with the insulin resistance and the metabolic syndrome. These observations are of particular interest because of the recognized relationship of FOXC2 haploinsufficiency to a variety of identified lymphedema syndromes. It is therefore attractive to conjecture that insulin resistance, perhaps mediated through polymorphisms of FOXC2,.confers secondary lymphedema risk and predisposes to the as yet poorly understood tendency for breast cancer survivors to acquire substantial, pathological deposits of adipose tissue in the affected extremities with chronicity of the lymphedema.

The specific aims of this proposal are as follows: (1) to quantitatively assess insulin sensitivity in late breast cancer survivors, equally divided among subjects who display clinical evidence of ipsilateral arm edema and those that do not; (2) to correlate the presence of relative insulin resistance to the expression of breast cancer-associated lymphedema. It is hypothesized that such an approach has the capability to lead to future elaboration of appropriate risk stratification and targeted therapeutic interventions; (3) as a pilot investigation, to sequence the FOXC2 gene, including the untranslated 5' region, in each these patients, to identify potential polymorphisms that might correlate both to the presence of insulin resistance and lymphedema risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the proposed studies must be survivors of breast cancer at a time point at least 4 years following the initial surgery and radiotherapy for the disease.
* Patients must have a history of unilateral axillary lymph node dissection.
* Patients referred to, or that receive their care within the Stanford University Breast Cancer Program and the Stanford Center for Lymphatic and Venous Disorders.
* Patients will be required to have the capacity to provide informed consent.

Exclusion Criteria:

* Patients with other serious systemic illness (renal failure, hepatic dysfunction, congestive heart failure, neurological or psychological impairment) that would confound the study or impair the patients' ability to participate.
* Patients will not be enrolled if they are taking drugs that affect carbohydrate metabolism.
* Patients with recurrent breast cancer or other forms of pre-existing lymphedema will be ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-07; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
assess insulin sensitivity in late breast cancer survivors | visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States